CLINICAL TRIAL: NCT04539288
Title: Pregnancy to Postpartum Transition of Serum Biomarkers in Women With Gestational Diabetes
Brief Title: Serum Biomarkers Associated With Postpartum T2DM in Women With GDM
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Dongyu Wang, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 50102013
Record Dates: First submitted 2018-09-05; First posted 2020-09-04 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Gestational Diabetes
Keywords: GDM; T2DM; NGT; lipids
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gestational diabetes mellitus: Women who were diagnosed GDM in 24-28 gestation weeks.

INTERVENTIONS:
Other:  — There is no intervention in this study.

SUMMARY:
Gestational diabetes mellitus (GDM) is commonly linked to the development of type 2 diabetes mellitus (T2DM). There is a need to characterize metabolic changes associated with GDM in order to find novel biomarkers for T2DM.

DETAILED DESCRIPTION:
GDM, a common complication of pregnancy, affects 17.8% of pregnancies worldwide per year. Women with a history of GDM have an approximately 7-fold higher risk for developing T2DM in the future than women without GDM. However, data on the factors associated with the development of T2DM in women with GDM are not widely available.

ELIGIBILITY:
Inclusion Criteria:

* Women who were dignosed GDM.
* Women with singleton pregnancy.
* Give birth in the First Affiliated Hospital in Sun Yat-sen University.

Exclusion Criteria:

* Women who were diagnosed PGDM.
* Younger than 18 years old.
* Older than 45 years old.
* Multiple pregnancy.
* Diagnosed DM before.
* Complicationg other diseases, like hypertension, thyroid diseases, etc.
* Taking any drug affect glucose and lipid metabolism.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: GDM Women.
Sampling Method: Probability Sample
Enrollment: 3099 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
T2DM | 4-6 weeks.
  Women with GDM develop T2DM in postpartum.

SECONDARY OUTCOMES:
IGT | 4-6 weeks.
  Women with GDM were impaired glucose intolerance in postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Dongyu Wang, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Obstetrics and Gynechology Department of the 1st affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China